CLINICAL TRIAL: NCT02550652
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Obinutuzumab in Patients With ISN/RPS 2003 Class III or IV Lupus Nephritis
Brief Title: A Study to Evaluate the Safety and Efficacy of Obinutuzumab Compared With Placebo in Participants With Lupus Nephritis (LN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA29748; 2015-002022-39 (EudraCT Number)
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; obinutuzumab; Methylprednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Obinutuzumab (Experimental): Participants will receive obinutuzumab 1000 milligrams (mg) intravenous (IV) infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose will be up titrated to a target dose of 2.0 - 2.5 grams per day (g/day) (or equivalent). Investigators, at their discretion, may use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants may receive 750-1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants will receive 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
  Interventions: Drug: Mycophenolate Mofetil/Mycophenolic Acid; Drug: Obinutuzumab; Drug: Methylprednisolone; Drug: Prednisone
- Placebo (Placebo Comparator): Participants will receive placebo matching to obinutuzumab IV infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose will be up titrated to a target dose of 2.0 - 2.5 g/day (or equivalent). Investigators, at their discretion, may use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants may receive 750-1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants will receive 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
  Interventions: Drug: Mycophenolate Mofetil/Mycophenolic Acid; Other: Placebo; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Mycophenolate Mofetil/Mycophenolic Acid — MMF/MPA will be administered as per schedule specified in the respective arm.
Drug: Obinutuzumab — Obinutuzumab will be administered as per schedule specified in the respective arm.
  Other Names: Gazyva, GA101, RO5072759
  Arms: Obinutuzumab
Other: Placebo — Placebo matching to obinutuzumab will be administered as per schedule specified in the respective arm.
  Arms: Placebo
Drug: Methylprednisolone — Methylprednisolone IV will be administered as per schedule specified in the respective arm.
Drug: Prednisone — Prednisone will be administered as per schedule specified in the respective arm.

SUMMARY:
This Phase II study will compare the efficacy and safety of obinutuzumab plus mycophenolate mofetil (MMF)/mycophenolic acid (MPA) with placebo plus MMF/MPA in participants with proliferative LN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Lupus Erythematosus (SLE), according to current American College of Rheumatology (ACR) criteria
* Diagnosis of International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV LN as evidenced by renal biopsy performed within 6 months prior to or during screening. Participants may co-exhibit Class V disease in addition to either Class III or Class IV disease
* Proteinuria (urine protein to creatinine ratio) greater than (>) 1.0
* For women who are not postmenopausal (greater than or equal to [>/=] 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 18 months after the last dose of study drug
* For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 12 months after the last dose of study drug and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* Retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia that is currently active and resulting from SLE
* Presence of rapidly progressive glomerulonephritis
* Severe renal impairment as defined by estimated Glomerular Filtration Rate (GFR) <30 milliliters per minute (mL/min) or the need for dialysis or renal transplant
* Greater than 50% of glomeruli with sclerosis on renal biopsy
* Treatment with cyclophosphamide or calcineurin inhibitors within the 3 months prior to randomization
* Unstable disease with thrombocytopenia or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies such as plasmapheresis or acute blood or platelet transfusions
* History of severe allergic or anaphylactic reactions to monoclonal antibodies or known hypersensitivity to any component of the obinutuzumab infusion
* Significant or uncontrolled medical disease in any organ system not related to SLE or LN, which, in the investigator's opinion, would preclude participant participation
* Concomitant chronic conditions, excluding SLE, (e.g., asthma, Crohn's disease) that required oral or systemic steroid use in the 52 weeks prior to screening
* Previous treatment with an anti-cluster of differentiation (CD20)-targeted therapy within 12 months
* Previous treatment with a biologic B-cell-targeted therapy (other than anti-CD20) within 6 months of randomization
* Known intolerance to MMF or MPA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (46):
- United States (7):
  - Univ of California, San Diego, La Jolla, California
  - Stanford University Medical Center, Palo Alto, California
  - Emory Uni ; Division of Rheumatology, Atlanta, Georgia
  - Suny Downstate Medical Center; Rheumatology, Brooklyn, New York
  - North Shore - Long Island Jewish Hospital Health System; Rheumatology & Allergy- Clinical Immunology, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University; Division of Nephrology, Columbus, Ohio
- Argentina (3):
  - Cemic; Haematology, Buenos Aires
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Organizacion Medica de Investigacion, San Nicolás
- Brazil (6):
  - Ser Servicos Especializados Em Reumatologia, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Instituto Scribner., Curitiba, Paraná
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Sao Paulo - UNIFES, São Paulo, São Paulo
- Colombia (4):
  - Clinica De La Costa, Barranquilla
  - Hospital Universitario San Ignacio, Bogotá
  - Riesgo De Fractura; Rheumatology, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- Hospital Clinica Catolica, Guadalupe, Costa Rica
- France (6):
  - HOPITAL HENRI MONDOR; SERVICE DE Nephrologie, Créteil
  - Hopital Claude Huriez; Internal Medicine, Lille
  - Hopital europeen Marseille; Service de medecine interne, Marseille
  - Groupe Hospitalier Pitie-Salpetriere; Service de Medecine Interne Ii, Paris
  - Hopital Bichat Claude Bernard; Nephrologie, Paris
  - Hopital Rangueil; Service de Nephrologie & D'Immunologie Clinique, Toulouse
- Israel (3):
  - Rambam Medical Center; Rheumatology, Haifa
  - Beilinson Medical Center; Rheumatology, Petah Tikva
  - Sheba Medical Center; Tel Hashomer, Ramat Gan
- Italy (2):
  - Ospedale San Giovanni Bosco; entro di Ricerche di Immunopatologia e Documentazione su Malattie Rare, Turin, Piedmont
  - Azienda Ospedaliera di Padova; Dipartimento di Medicina - UOC di Reumatologia, Padua, Veneto
- Mexico (7):
  - Unidad de Reumatologia Rehabilitacion Integral; Centro Medico Del Angel, Mexicali, Estado de Baja California
  - Unidad de Investigacion en Enfermedades Cronico-Degenerativa; Reumatologia, Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Basica Y Clinica S.C.; Reumatologia, Guadalajara, Jalisco
  - Hospital General De Mexico; Rheumatology, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Ciencias Médicas Y de La Nutricion Zubirán, Mexico City, Mexico CITY (federal District)
  - Centro de Investigación Clínica de Morelia S.C., Morelia, Michoacán
  - Centro de Investigación de Tratamientos Innovadores de Sinaloa (CITI), Culiacán, Sinaloa
- Trial Labs, Panama City, Panama
- Peru (4):
  - Instituto de Ginecología y Reproducción, Lima
  - Centro de Investigación Delgado; Clinica Delgado, Miraflores
  - Centro de Investigaciones Medicas/Hospital Maria Auxiliadora, San Juán de Miraflores
  - Hospital Nacional Cayetano Heredia; Rheumatology, San Martín de Porres
- Spain (2):
  - Hospital Clinic i Provincial; Servicio de Nefrologia, Barcelona
  - Hospital Regional Universitario Carlos Haya; Servicio de Reumatologia, Málaga

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Rovin BH, Furie RA, Ross Terres JA, Giang S, Schindler T, Turchetta A, Garg JP, Pendergraft WF 3rd, Malvar A. Kidney Outcomes and Preservation of Kidney Function With Obinutuzumab in Patients With Lupus Nephritis: A Post Hoc Analysis of the NOBILITY Trial. Arthritis Rheumatol. 2024 Feb;76(2):247-254. doi: 10.1002/art.42734. Epub 2023 Nov 10. PMID 37947366
- [Derived] Furie RA, Aroca G, Cascino MD, Garg JP, Rovin BH, Alvarez A, Fragoso-Loyo H, Zuta-Santillan E, Schindler T, Brunetta P, Looney CM, Hassan I, Malvar A. B-cell depletion with obinutuzumab for the treatment of proliferative lupus nephritis: a randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2022 Jan;81(1):100-107. doi: 10.1136/annrheumdis-2021-220920. Epub 2021 Oct 6. PMID 34615636
- [Derived] Dossier C, Hogan J. Response to Majeranowski. Pediatr Nephrol. 2021 Jun;36(6):1653. doi: 10.1007/s00467-021-04982-4. Epub 2021 Mar 10. No abstract available. PMID 33693991

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 126 patients were enrolled in the study however one patient randomized to obinutuzumab did not receive study treatment due to a positive pregnancy test, but prior to the first study drug infusion; therefore a total of 125 patients are included in the analysis.
Groups:
- OBINUTUZUMAB 1000MG and MMF: Participants received obinutuzumab 1000 milligrams (mg) intravenous (IV) infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose was up titrated to a target dose of 2.0 - 2.5 grams per day (g/day) (or equivalent). Investigators, at their discretion, could use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants could receive 1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants received 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
- PLACEBO and MMF: Participants received placebo matching to obinutuzumab IV infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose was up titrated to a target dose of 2.0 - 2.5 g/day (or equivalent). Investigators, at their discretion, could use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants could receive 1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants received 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
Period: Overall Study
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Started | 63 | 62
Completed | 55 | 44
Not Completed | 8 | 18
Not completed — Death | 1 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Post Trial Access | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Receipt of additional therapies that reduce peripheral B cell counts | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.1 (9.8) | 31.9 (10.1) | 32.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Or Latino | 42 | 49 | 91
  Not Hispanic Or Latino | 20 | 12 | 32
  Not Stated | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 17 | 28
  Asian | 3 | 2 | 5
  Black or African American | 6 | 5 | 11
  Multiple | 1 | 0 | 1
  Native Hawaiian or other Pacific Islande | 1 | 0 | 1
  Unknown | 13 | 12 | 25
  White | 28 | 26 | 54
Circulating CD19-Positive B-Cell Levels [Mean (Standard Deviation); unit: cells/uL] — Population: The number analyzed indicates the number of participants with non-missing results at baseline. Values below the level of quantification have been excluded from the analysis.
  cells/uL
    number analyzed (Participants) | 48 | 48 | 96
    (all) | 328 (331) | 353 (454) | 341 (395)
Region of Enrollment [Count of Participants; unit: Participants] — Population: The number analyzed represents the number of patients contributing to summary statistics.
  Participants
    number analyzed (Participants) | 62 | 61 | 123
    Asia | 2 | 2 | 4
    European Union | 16 | 5 | 21
    Latin America | 37 | 46 | 83
    United States | 7 | 8 | 15
Lupus Nephritis (LN) Biopsy Class [Number; unit: Participants] — Participants were graded as Class III or Class IV using the classification by the International Society of Nephrology and the Renal Pathology Society (ISN/RPS):
  Class III Focal LN (< 50% of glomeruli) III (A): active lesions III (A/C): active and chronic lesions III (C): chronic lesions
  Class IV Diffuse LN (≥50% glomeruli) Diffuse segmental (IV-S) or global (IV-G) LN IV (A): active lesions IV (A/C): active and chronic lesions IV (C): chronic lesions Stage IV is considered to have worse clinical outcome than stage III.
  Participants
    III | 14 | 17 | 31
    IV | 49 | 45 | 94
Urine Protein Creatinine Ratio (UPCR) [Mean (Standard Deviation); unit: mg/mg] — Population: Due to a central lab error, uPCR was not available for the first 5 patients at baseline
  mg/mg
    number analyzed (Participants) | 60 | 60 | 120
    (all) | 3.32 (2.66) | 2.93 (2.46) | 3.12 (2.56)
Serum creatinine [Mean (Standard Deviation); unit: (mg/dL)] | 0.87 (0.34) | 0.8 (0.32) | 0.84 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Protocol Defined Complete Renal Response (CRR) at Week 52
Description: Percentage of participants with normalization of serum creatinine, inactive urinary sediment (as evidenced by < 10 red blood cells (RBCs)/high-power field (HPF) and the absence of red cell casts) and urinary protein to creatinine ratio < 0.5. Normalization of serum creatinine is defined as serum creatinine ≤ the upper limit of normal (ULN) range of central laboratory values if baseline (Day 1) serum creatinine is above the ULN or serum creatinine ≤ 15% above baseline and ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine is above the ULN range of central laboratory values.
Time Frame: From baseline to Week 52
Population: Modified intent-to-treat population will include all randomized participants who have received any amount of study drug. Participants who received an incorrect therapy were reported under the treatment arm to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 22 | 14
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.1145, Cochran-Mantel-Haenszel — Stratified by race (Afro Caribbean/African American vs. Others) and region (US vs. non-US sites). Statistically significant at pre-specified alpha of 20%; Difference in Percentage of Participants = 12.3, 95% CI 2-sided [-3.4 to 28.1]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.1145, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants; Difference in Percentage of Participants = 12.3, 80% CI 2-sided [2.1 to 22.6]

2. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined Overall Response (OR) at Week 52
Description: OR includes both CRR and partial renal response (PRR). CRR as defined in the primary outcome measure above. PRR defined as 50% improvement in urine protein:creatinine ratio, with one of following conditions met: 1. If baseline urine protein:creatinine ratio is ≤ 3.0, then urine protein:creatinine ratio of <1.0. 2. If baseline protein:creatinine ratio is > 3.0, then urine protein:creatinine ratio of <3.0, serum creatinine ≤15% above baseline value, and no urinary red cell casts and either RBCs/HPF ≤50% above baseline or <10 RBCs/HPF.
Time Frame: From baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 35 | 22
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0246, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 20.1, 95% CI [3.0 to 37.2]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0246, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 20.1, 80% CI 2-sided [8.9 to 31.3]

3. Secondary Outcome: Time to OR Over 52 Weeks
Description: OR includes both CRR and partial renal response(PRR). CRR as defined in the primary outcome measure above. PRR defined as 50% improvement in upcr, with one of these conditions met: 1. If baseline upcr is ≤3.0, then upcr of <1.0. 2. If baseline pcr is > 3.0, then upcr of <3.0, serum creatinine ≤15% above baseline value, and no urinary red cell casts and either RBCs/HPF ≤50% above baseline or <10 RBCs/HPF. Percentage of participants with response at various time points were measured using Kaplan Meier method.
Time Frame: From baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants
  Week 12 | 55 | 59
  Week 24 | 33 | 37
  Week 36 | 21 | 29
  Week 52 | 14 | 21
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0744, Log Rank

4. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined Partial Renal Response (PRR) at Week 52
Description: PRR defined as serum creatinine ≤15% above baseline value, no urinary red cell casts and either RBCs/HPF ≤ 50% above baseline or < 10 RBCs/HPF, 50% improvement in urine protein:creatinine ratio, with one of following conditions met: 1. If baseline urine protein:creatinine ratio is ≤ 3.0, then a urine protein:creatinine ratio of < 1.0. 2. If baseline protein:creatinine ratio is > 3.0, then a urine protein:creatinine ratio of < 3.0.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 35 | 21
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0150, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 21.7, 95% CI [4.7 to 38.7]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0150, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 21.7, 80% CI 2-sided [10.6 to 32.8]

5. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined CRR at Week 24
Description: CRR defined as normalization of serum creatinine, inactive urinary sediment (as evidenced by < 10 red blood cells (RBCs)/high-power field (HPF) and the absence of red cell casts) and urinary protein to creatinine ratio < 0.5. Normalization of serum creatinine is defined as serum creatinine ≤ the upper limit of normal (ULN) range of central laboratory values if baseline (Day 1) serum creatinine is above the ULN or serum creatinine ≤ 15% above baseline and ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine is ≤ the ULN range of central laboratory values.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 16 | 17
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.8461, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -2.0, 95% CI 2-sided [-17.5 to 13.4]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.8461, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = -2.0, 80% CI 2-sided [-12.1 to 8.1]

6. Secondary Outcome: Time to CRR Over 52 Weeks
Description: CRR included normalization of serum creatinine, inactive urinary sediment (as evidenced by < 10 RBCs/HPF and the absence of red cell casts) and urinary protein to creatinine ratio < 0.5. Normalization of serum creatinine is defined as serum creatinine ≤ the ULN range of central laboratory values if baseline serum creatinine is above the ULN or serum creatinine ≤ 15% above baseline and ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine is ≤ the ULN range of central laboratory values. Percentage of participants with response at various time points were measured using Kaplan Meier method.
Time Frame: From Baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants
  Week 12 | 61 | 60
  Week 24 | 47 | 48
  Week 36 | 38 | 38
  Week 52 | 27 | 33
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.3530, Log Rank

7. Secondary Outcome: Change From Baseline in Anti-Double Stranded Deoxyribonucleic Acid (Anti-dsDNA) Antibody Levels at Week 52
Description: Anti-dsDNA antibodies are a group of anti-nuclear autoantibodies targeting double stranded DNA.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
log IU/mL | -0.810 (1.054) | -0.076 (1.103)
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in Adjusted Mean = -0.81, 95% CI 2-sided [-1.13 to -0.491]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in Adjusted Mean = -0.81, 80% CI 2-sided [-1.019 to -0.602]

8. Secondary Outcome: Change From Baseline in Complement Component 3 (C3) Levels at Week 52
Description: Complement C3 is a blood test that reflects activation of complement pathway associated with immune deposition in certain autoimmune diseases.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
g/L | 0.311 (0.302) | 0.106 (0.273)
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0004, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in Adjusted Mean = 0.178, 95% CI 2-sided [0.081 to 0.275]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0004, ANCOVA; Difference in Adjusted Mean = 0.178, 80% CI 2-sided [0.115 to 0.241]

9. Secondary Outcome: Change From Baseline in C4 Levels at Week 52
Description: Complement C4 is a blood test that reflects activation of complement pathway associated with immune deposition in certain autoimmune diseases.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
g/L | 0.101 (0.117) | 0.004 (0.164)
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p < 0.0001, ANCOVA; Stratified by race (Afro Caribbean/African American vs. Others) and region (US vs. non-US sites); Difference in Adjusted Mean = 0.088, 95% CI [0.052 to 0.124]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in Adjusted Mean = 0.088, 80% CI 2-sided [0.065 to 0.112]

10. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined Modified CRR (mCRR1) at Week 52
Description: mCRR1 has got two components only, i.e. serum Creatinine and urinary protein to creatinine ratio. mCRR1 is defined by attainment of normalization of serum creatinine as evidenced by 1.) serum creatinine ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine is above the ULN or serum creatinine ≤15% above baseline and ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine ≤ the ULN range of central laboratory values and 2.) Urinary protein to creatinine ratio <0.5.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 25 | 16
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0900, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 13.9, 95% CI [-2.4 to 30.1]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.0900, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 13.9, 80% CI 2-sided [3.2 to 24.5]

11. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined Second mCRR (mCRR2) at Week 52
Description: mCRR2 is defined by normalization of serum creatinine, inactive urinary sediment (as evidenced by < 10 RBCs/HPF and the absence of red cell casts), and urinary protein to creatinine ratio <0.5. Normalization of serum creatinine as evidenced by the following: Serum creatinine ≤15% above baseline if baseline (Day 1) serum creatinine is above the normal range of the central laboratory values or ≤ the ULN range of central laboratory values if baseline (Day 1) serum creatinine is ≤ the ULN range of central laboratory values.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 28 | 21
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.1838, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 10.6, 95% CI 2-sided [-6.4 to 27.6]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.1838, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 10.6, 80% CI 2-sided [-0.5 to 21.7]

12. Secondary Outcome: Percentage of Participants Who Achieve Protocol Defined Third mCRR (mCRR3) at Week 52
Description: mCRR3 is defined by normalization of serum creatine as evidenced by serum creatinine ≤ the ULN range of central laboratory values and urinary protein to creatinine ratio < 0.5.
Time Frame: Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Participants | 29 | 24
Statistical Analysis 1: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.3726, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 7.3, 95% CI 2-sided [-10.0 to 24.6]
Statistical Analysis 2: Comparison: OBINUTUZUMAB 1000MG and MMF vs PLACEBO and MMF; Test type: Superiority; p = 0.3726, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Percentage of Participants = 7.3, 80% CI 2-sided [-4.0 to 18.6]

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs, including AEs of Special Interest were reported based on the national cancer institute common terminology criteria for AEs, Version 4.0 (NCI-CTCAE, v4.0). Reported are the number of subjects with AEs, Grade 3-5 AEs, and Serious Adverse Events (SAEs), Infections and Serious infections. The AEs reported do not include events after the receipt of rescue medications.
Time Frame: From baseline to approximately 7 years and 8 months
Population: The safety population was defined as all participants who have received any amount of study medication. Participants are reported under the therapy they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 64 | 61
Participants
  Adverse Events | 58 | 54
  Grade 3 AEs | 19 | 15
  Grade 4 AEs | 6 | 7
  Grade 5 AEs | 1 | 2
  Serious Adverse Events | 16 | 17
  Infections | 48 | 38
  Serious infections | 5 | 10

14. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest: Infusion Related Reactions, Grade 3 or Higher Infections, Drug-related Neutropenia and Drug-related Thrombocytopenia
Description: Infusion related reaction is defined as any event reported within 24 hours of infusion and thought to be causally related to the investigational agent by the investigator. Grade 3 or higher infections include all events of Grade 3 to 5 under the SOC of infections and infestations. Drug-related neutropenia is defined as events in the Roche AE Grouped Term (AEGT) "Neutropenia and associated complications" and thought to be causally related to the investigational agent by the investigator. Drug-related thrombocytopenia is defined as events in the Standard MedDRA Query (SMQ) "Haematopoietic Thrombocytopenia narrow" and thought to be causally related to the investigational agent by the investigator.
Time Frame: From baseline to approximately 7 years and 8 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 64 | 61
Participants
  Infusion Related Reactions | 10 | 6
  Grade 3 or Higher Infections | 4 | 11
  Drug-related Neutropenia | 3 | 2
  Drug-related Thrombocytopenia | 0 | 0

15. Secondary Outcome: Percentage of Participants With Anti-Drug Antibody (ADA) to Obinutuzumab
Description: Antibodies are a blood protein produced in response to and counteracting a specific antigen.
Time Frame: From baseline to approximately 7 years and 8 months
Population: Pharmacokinetic population included all patients randomized to and received any dose of obinutuzumab given as study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 63
Participants | 7

16. Secondary Outcome: Percent Change From Baseline in Circulating CD19-Positive B-Cell Levels
Description: CD19+ B cell is a B-lymphocyte with a transmembrane protein that is encoded by the gene CD19.
Time Frame: Baseline, Week 2, Week 4, Week 12, Week 24, Week 52, Week 104, B Cell Follow-Up (Bcfu) at months 6, 12, 18, 24, 30, 36, 42 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change of cells/uL
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
Percent change of cells/uL
  Week 2: number analyzed (Participants) | 39 | 42
  Week 2 | -97.469 (12.899) | 39.293 (145.247)
  Week 4: number analyzed (Participants) | 45 | 36
  Week 4 | -98.777 (5.235) | -5.186 (78.469)
  Week 12: number analyzed (Participants) | 41 | 45
  Week 12 | -97.045 (15.506) | 0.661 (134.421)
  Week 24: number analyzed (Participants) | 42 | 37
  Week 24 | -96.628 (10.207) | -11.446 (86.793)
  Week 52: number analyzed (Participants) | 39 | 42
  Week 52 | -98.620 (5.677) | 37.695 (220.857)
  Week 104: number analyzed (Participants) | 5 | 2
  Week 104 | 77.123 (380.111) | -76.055 (31.519)
  Bcfu Month 6: number analyzed (Participants) | 13 | 5
  Bcfu Month 6 | 105.043 (402.281) | -73.889 (19.755)
  Bcfu Month 12: number analyzed (Participants) | 5 | 2
  Bcfu Month 12 | 77.123 (380.111) | -76.055 (31.519)
  Bcfu Month 18: number analyzed (Participants) | 3 | 1
  Bcfu Month 18 | -83.159 (16.701) | -11.418 (NA) — The standard deviation could not be derived from the data of 1 participant.
  Bcfu Month 24: number analyzed (Participants) | 2 | 0
  Bcfu Month 24 | -93.603 (8.836) |
  Bcfu Month 30: number analyzed (Participants) | 3 | 0
  Bcfu Month 30 | -59.950 (50.807) |
  Bcfu Month 36: number analyzed (Participants) | 2 | 0
  Bcfu Month 36 | -99.163 (0.973) |
  Bcfu Month 42: number analyzed (Participants) | 1 | 0
  Bcfu Month 42 | -99.084 (NA) — The standard deviation could not be derived from the data of 1 participant. |
  Bcfu Month 48: number analyzed (Participants) | 1 | 0
  Bcfu Month 48 | -99.851 (NA) — The standard deviation could not be derived from the data of 1 participant. |

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Obinutuzumab
Time Frame: Week 0, Week 24, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 63
ug/mL
  Week 0-24 | 559 (112)
  Week 24-52 | 605 (115)
  Week 0-52 | 605 (115)

18. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Obinutuzumab
Time Frame: Baseline to Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ug/mL*day
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 63
ug/mL*day
  Week 0-24 | 10595 (4016)
  Week 24-52 | 15811 (5543)
  Week 0-52 | 26406 (9027)

19. Secondary Outcome: Systemic Clearance of Obinutuzumab
Time Frame: Day 0, Week 24, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 63
L/day
  Day 0 | 0.255 (0.136)
  Week 24 | 0.147 (0.0564)
  Week 52 | 0.137 (0.0535)

20. Secondary Outcome: Volume of Distribution Under Steady State (Vss) of Obinutuzumab
Time Frame: Day 0, Week 24, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Litre (L)
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 63
Litre (L)
  Day 0 | 3.67 (0.591)
  Week 24 | 3.67 (0.591)
  Week 52 | 3.67 (0.591)

21. Secondary Outcome: Terminal Plasma Half-Life (t1/2) of Obinutuzumab
Time Frame: Day 0, Week 24, Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: day
Arm/Group | OBINUTUZUMAB 1000MG and MMF
Number analyzed (Participants) | 64
day
  Day 0 | 13.1 (3.7)
  Week 24 | 20.5 (5.6)
  Week 52 | 22.1 (6.7)

22. Secondary Outcome: Change From Baseline of Participant's Global Assessment of Disease Activity Visual Analog Scale (VAS) Score
Description: Each VAS had a range from 0-100 with higher scores indicating greater symptom impact on global health status.
Time Frame: Baseline (Day 1), Weeks 4, 12, 24, 36, 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | OBINUTUZUMAB 1000MG and MMF | PLACEBO and MMF
Number analyzed (Participants) | 63 | 62
score on scale
  Baseline: number analyzed (Participants) | 58 | 60
  Baseline | 41.3 (25.59) | 39.4 (24.76)
  Week 4: number analyzed (Participants) | 55 | 57
  Week 4 | -14.4 (18.28) | -8.7 (22.69)
  Week 12: number analyzed (Participants) | 57 | 60
  Week 12 | -19.9 (25.07) | -11.6 (25.22)
  Week 24: number analyzed (Participants) | 54 | 56
  Week 24 | -25.0 (25.17) | -20.8 (24.74)
  Week 36: number analyzed (Participants) | 54 | 57
  Week 36 | -24.8 (25.71) | -19.6 (25.04)
  Week 52: number analyzed (Participants) | 54 | 56
  Week 52 | -25.4 (26.49) | -23.3 (25.76)

ADVERSE EVENTS:
Time Frame: From baseline to approximately 7 years and 8 months
Description: The safety population was defined as all participants who have received any amount of study medication.
Groups:
- OBINUTUZUMAB 1000MG + MMF: Participants received obinutuzumab 1000 milligrams (mg) intravenous (IV) infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose was up titrated to a target dose of 2.0 - 2.5 grams per day (g/day) (or equivalent). Investigators, at their discretion, could use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants could receive 1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants received 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
- PLACEBO + MMF: Participants received placebo matching to obinutuzumab IV infusion on Days 1, 15, 168, and 182 along with MMF/MPA at a starting dose of 1500 mg/day (or equivalent) administered orally in 2 or 3 divided doses. MMF/MPA dose was up titrated to a target dose of 2.0 - 2.5 g/day (or equivalent). Investigators, at their discretion, could use MPA as a substitute for MMF, with a 360 mg dose being equivalent to a 500 mg dose of MMF. During screening or at randomization, if clinically indicated, participants could receive 1000 mg methylprednisolone IV once daily for up to 3 days to treat underlying LN clinical activity. Participants received 0.5 mg/kg oral prednisone, tapering this prednisone dose, per protocol, starting on Day 16 and reducing the prednisone dosage to 7.5 mg/day by Week 12.
Arm/Group | OBINUTUZUMAB 1000MG + MMF | PLACEBO + MMF
All-Cause Mortality (participants affected / at risk) | 1/64 | 4/61
Serious Adverse Events (participants affected / at risk) | 17/64 | 18/61
Other Adverse Events (participants affected / at risk) | 51/64 | 39/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBINUTUZUMAB 1000MG + MMF (N=64) | PLACEBO + MMF (N=61)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 1 (2)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS CHORIORETINITIS (Infections and infestations) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS MYOCARDITIS (Infections and infestations) | 0 (0) | 1 (1)
DISSEMINATED CYTOMEGALOVIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ENDOMETRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 3 (3)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
IDIOPATHIC INTRACRANIAL HYPERTENSION (Nervous system disorders) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
LUPUS NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
INTUSSUSCEPTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (2)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1)
MYELITIS TRANSVERSE (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Infections and infestations) | 1 (1) | 0 (0)
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OBINUTUZUMAB 1000MG + MMF (N=64) | PLACEBO + MMF (N=61)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 4 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (7) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 6 (7) | 3 (3)
CHEST PAIN (General disorders) | 0 (0) | 4 (4)
BRONCHITIS (Infections and infestations) | 13 (15) | 5 (8)
CONJUNCTIVITIS (Infections and infestations) | 4 (6) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 3 (4) | 6 (9)
HERPES ZOSTER (Infections and infestations) | 5 (6) | 6 (7)
INFLUENZA (Infections and infestations) | 4 (4) | 2 (3)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 6 (8)
PHARYNGITIS (Infections and infestations) | 5 (8) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (8) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 14 (19) | 12 (20)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 7 (7) | 6 (7)
HEADACHE (Nervous system disorders) | 5 (7) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 4 (4)
HYPERTENSION (Vascular disorders) | 6 (6) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (5)
INSOMNIA (Psychiatric disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT02550652/Prot_004.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT02550652/SAP_005.pdf